CLINICAL TRIAL: NCT03922009
Title: The Effect of Virtual Reality on Patients With Anxiety Over Surgeries Under Spinal Anesthesia-A Case Study of Orthopedic Lower Limb Surgery
Brief Title: The Effect of Virtual Reality on Patients With Anxiety Over Surgeries Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University Hospital (Other)
Responsible Party: Principal Investigator, YANG,HSIN-CHIEH, National Yang-Ming University Hospital, National Yang Ming Chiao Tung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NYMUH-IRB No.2018A015
Record Dates: First submitted 2019-01-19; First posted 2019-04-19 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Virtual Reality
Keywords: Virtual Reality；Anxiety

STUDY DESIGN:
Intervention Model Description: 50 people in the control group 50 people in the experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality group (Experimental): The primary objective of this study was to evaluate the use of VR to reduce anxiety in spinal anesthesia patients compared with controls
  Interventions: Device: Virtual Reality
- control group (No Intervention): General routine care

INTERVENTIONS:
Device: Virtual Reality — The primary objective of this study was to evaluate the use of VR to reduce anxiety in spinal anesthesia patients compared with controls
  Arms: Virtual Reality group

SUMMARY:
The main purposes of this study are as follows:

First, to understand the effect of virtual reality on the subjective feelings of anxiety in patients with orthopaedic lower limb surgery for spinal anesthesia.

Second, to understand the effects of virtual reality on the systolic blood pressure, diastolic blood pressure, mean arterial pressure, heartbeat, respiration and other physiological parameters in the operation of orthopedic lower extremity surgery patients with spinal anesthesia.

Third, to understand the effect of using virtual reality in surgery to reduce the use of sedative drugs and the degree of pain in patients with orthopedic lower extremity surgery.

DETAILED DESCRIPTION:
Surgery is a serious source of stress for the general patient and can increase the patient's anxiety. which is It is normal to show obvious anxiety in patients undergoing surgery, but if the degree of anxiety is serious, it may lead Negative physiological manifestations, such as slow wound healing, increase the risk of infection and may affect the induction of anesthesia It requires more anesthesia dose during surgery, which hinders recovery time. Most studies have confirmed surgery Playing music in the room can alleviate the anxiety and pain of the patients, but the music preference is subjective and some people like it.

There must be people who hate it, and the operating room is not a quiet space. There are many sound sources in the operating room., such as the sound of surgical instruments, the warning sound of physiological monitors, the voice of the staff, these It will be a source of anxiety for patients. Instrument noise averages up to 60 decibels, including neurosurgery, orthopedics It can even exceed 100 decibels. Foreign scholars believe that playing music at this time will only aggravate the noisy environment.The attention of the staff. Therefore, it is hoped that by using virtual reality to provide images and sounds during surgery, hijacking The patient's auditory, visual, and proprioception creates an immersive, distracting approach that reduces the cause of the ring Anxiety brought by the environment helps spinal anesthesia patients to reduce anxiety during surgery and increase psychological comfort To reduce the use of sedative drugs during surgery.

ELIGIBILITY:
Inclusion Criteria:

1. population: acceptance of lower extremity fractures in patients with spinal anesthesia.
2. Anesthesia classification (ASA): I-III.
3. Age: 20 years old to 70 years of age.

Exclusion Criteria:

1. Mental illness and taking related drugs.
2. Visually impaired and hearing impaired.
3. Being unable to communicate or illiterate.
4. The condition changes or is critical, and the intensive care unit is admitted after the operation.
5. Contact isolation.
6. Trauma of the head and wounds on the head.
7. History of motion sickness and vertigo.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Anxiety | After anesthesia until the end of surgery(intraoperative )
  First, to understand the effect of virtual reality on the subjective feelings of anxiety in patients with orthopaedic lower limb surgery for spinal anesthesia.USE State-Trait Anxiety Inventory；STAI

SECONDARY OUTCOMES:
physiological parameters | After anesthesia until the end of surgery(intraoperative )
  Second, to understand the effects of virtual reality on the mean arterial pressure physiological parameters in the operation of orthopedic lower extremity surgery patients with spinal anesthesia.
physiological parameters | After anesthesia until the end of surgery(intraoperative )
  Second, to understand the effects of virtual reality on the heartbeat physiological parameters in the operation of orthopedic lower extremity surgery patients with spinal anesthesia.
physiological parameters | After anesthesia until the end of surgery(intraoperative )
  Second, to understand the effects of virtual reality on the respiration physiological parameters in the operation of orthopedic lower extremity surgery patients with spinal anesthesia.

OTHER OUTCOMES:
sedative drugs | After anesthesia until the end of surgery(intraoperative )
  Third, to understand the effect of using virtual reality in surgery to reduce the use of sedative drugs and the degree of pain in patients with orthopedic lower extremity surgery.USE Numerical Rating Scale；NRS

CONTACTS AND LOCATIONS:
Overall Officials: HSIN-CHIEH YANG, Bachelor, Principal Investigator — National Yang Ming Chiao Tung University Hospital
Locations (1):
- National Yang-Ming University Hospital, Yilan, Yilan County, Taiwan

IPD SHARING:
Plan to Share IPD: No